CLINICAL TRIAL: NCT03630549
Title: Village-based Refill of ART After Same-day ART Start vs Clinic-based ART Refill for HIV-positive Individuals Not on ART During Home-based HIV Testing (Part B of GET ON Research Project)
Brief Title: Village-based vs Clinic-based ART Care - a Cluster Randomized Controlled Trial in Lesotho
Acronym: VIBRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niklaus Labhardt (Other)
Collaborators: Ministry of Health, Lesotho (Other Government); SolidarMed (Other); University of Basel (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Niklaus Labhardt, Principal Investigator, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VIBRA
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS
Keywords: HIV; Village Health Worker; Differentiated Care; Lesotho; Africa; antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): 1. Offer of home-based same-day ART initiation
  2. Clinic-based ART visit/refill Who: Nurse Where: Nurse-led health facility When: Follow-up interval of max. 3 months What: TB screening, Screening for other opportunistic infections, Screening for ART-related toxicities, adherence assessment, assessment whether patient visited any medical facility since last appointment, addressing basic psychosocial problems, ART (+CTX/IPT) dispensing
  3. No SMS intervention
  Interventions: Other: Standard of Care
- Village-based ART refill (Experimental): 1. Offer of home-based same-day ART initiation
  2. Offer of Village-based ART visit/refill Who: VHW Where: At VHW's home* When: Follow-up interval of max. 3 months What: TB screening, Screening for other opportunistic infections, Screening for ART-related toxicities, adherence assessment, assessment whether patient visited any medical facility since last appointment, addressing basic psychosocial problems, ART (+CTX/IPT) dispensing
     *Except at 6 and 12 months follow-up: visit at health facility for laboratory assessment (viral load)
  3. Offer of Individually customized SMS
     * Monthly reminder SMS: to pick up ART
     * SMS communicating VL result
  Interventions: Other: Village-based ART refill

INTERVENTIONS:
Other: Standard of Care — Clinic-based HIV care
  Arms: Standard of Care
Other: Village-based ART refill — Option to get ART refill and care by the village health worker
  Other Names: VIBRA
  Arms: Village-based ART refill

SUMMARY:
This cluster-randomized trial tests a differentiated care model for HIV-positive individuals not on ART during a home-based HIV testing campaign in rural Lesotho, Southern Africa. In intervention clusters, patients are offered a differentiated ART delivery package with two features. Firstly, drug-refill and follow-up are provided by village health workers (VHW), reducing clinic visits to twice a year for laboratory assessment. Secondly, participants have the option of receiving individually tailored adherence reminders and viral load result notifications via SMS.

DETAILED DESCRIPTION:
The VIBRA trial is a cluster randomized controlled, open-label, superiority trial in a resource-limited setting. The trial is linked to a another trial, the HOSENG (HOme-based SElf-testiNG) trial, that is described elsewhere (NCT03598686). Together, they consitute the GET ON (GETing tOwards Ninety) research project. The HOSENG study, with its home-based HIV testing campaign, provides the recruitment platform for the VIBRA study. The reasons for this interlinked design are: a) potential study participants for VIBRA trial (HIV-positive individuals not on ART) are to be recruited during a home-based HIV testing campaign and hence, it allows us to assess the entire HIV care cascade in one larger project, and b) both trials rely on interventions involving VHWs, who need to be randomized and specifically trained. Therefore, it is efficient and feasible to run both trials parallel and randomize at one time point only. The rational for a cluster randomized design is the reliance of the trial on the VHWs and, thus, the high risk of cross-contamination between the study arms if randomization would be done at individual level.

ELIGIBILITY:
Inclusion Criteria for clusters:

* the cluster is clearly confined to the catchment area of one of the study clinics
* the cluster has at least one registered VHW who is willing to participate and fulfills the following criteria:
* is at least 18 years of age
* has adequate reading and writing skills
* successfully passes the training assessment
* village authority (village chief) is willing to participate in trial

Exclusion criteria for clusters:

* Village authority (=village chief) opposed to trial participation (verbal assent)
* Village health worker opposed to trial participation or not fulfilling the minimum requirements mentioned above

Inclusion Criteria for individuals:

* Individual is a household member of the visited households of the respective clusters
* Individual is confirmed HIV-positive
* Individual has never taken ART (ART-naïve) or has stopped ART more than 30 days prior (ART-defaulters)
* Individual is ≥10 years old and has a body weight of ≥35kg
* Individual is not in care for high blood pressure or diabetes (high blood sugar)
* HIV-positive individual wishes to get care outside the study districts

Exclusion criteria individuals:

* The household member is absent at the time of the campaign
* HIV-positive individual is taking ART or stopped less than 30 days ago
* HIV-positive individual is physically, mentally, or emotionally not able to participate in the study, in the opinion of the investigators or study staff
* HIV-positive individual is in care for high blood pressure (hypertension) or high blood sugar (diabetes) - proof of documentation or medication needed
* HIV-positive individual wishes to get care outside the study districts

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
12-months viral suppression | 12 months (range: 10 - 15 months) after enrolment.
  Viral suppression at 12 months, defined as the proportion of all participants with a VL <20 copies/mL
12-months viral suppression (<400copies/mL) | 12 months (range: 10 - 15 months) after enrolment.
  Viral suppression at 12 months, defined as the proportion of all participants with a VL <400 copies/mL

SECONDARY OUTCOMES:
6-months viral suppression | 6 months (range 5 - 8 months) after enrolment
  Viral suppression at 6 months, defined as the proportion of all participants with a VL <20 copies/mL
Alternative viral suppression at 12 months | 12 months (range 10 - 15 months) after enrolment.
  The proportion of all participants with a VL <1000 copies/mL
Alternative viral suppression at 6 months | 6 months (range 5 - 8 months) after enrolment
  The proportion of all participants with a VL <1000 copies/mL
Sustained viral suppression | 12 months (range 5 - 15 months) after enrollment
  The proportion of all participants with a VL <20 copies/mL at 6 (range 5 - 8 months) as well as at 12 months (range 10 - 15 months) after enrolment
1-month linkage to care | 30 days after enrollment
  Linkage to care within 1 month, defined as the proportion of all participants attending the first clinic- or VHW-based ART visit at least once within 1 month after enrolment
3-months linkage to care | 90 days
  Linkage to care within 3 months, defined as the proportion of all participants attending the first clinic- or VHW-based ART visit at least once within 3 months after enrolment
6-months retention in care | 5-8 months after enrollment
  The proportion of all participants active in care at a health facility or at the VHW 6 months (range 5 - 8 months) after enrollment
12-months retention in care | 12 months (range 10 - 15 months) after enrolment
  the proportion of all participants active in care at a health facility or at the VHW
All-cause mortality at 12 months | 12 months (range 10 - 15 months) after enrolment
  The proportion of all participants who died
Loss to follow-up at 12 months | 12 months (range 10 - 15 months) after enrollment
  The proportion of all participants lost to follow-up
Confirmed transfer out at 12 months | 12 months (range 10 - 15 months) after enrolment
  The proportion of all participants who transferred out to any other health facility (than the one initially registered) outside the study districts with a proof of transfer (documented proof of follow-up visit or laboratory test)
Unconfirmed transfer out at 12 months | 12 months (range 10 - 15 months) after enrolment
  The proportion of all participants who transferred out to any other health facility (than the one initially registered) outside the study districts without a proof of transfer at 12 months (range 10 - 15 months) after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus D Labhardt, MD, Principal Investigator — University Hospital Basel & Swiss Tropical and Public Health Institute; Tracy R Glass, PhD, Study Chair — Swiss Tropical & Public Health Institute; Manuel Battegay, MD, Study Chair — University Hospital, Basel, Switzerland; Josephine Muhairwe, MD, Study Chair — SolidarMed - Swiss Organization for Health in Africa
Locations (2):
- Lesotho (2):
  - District of Butha-Buthe, Butha-Buthe
  - District of Mokhotlong, Mokhotlong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amstutz A, Lejone TI, Khesa L, Kopo M, Kao M, Muhairwe J, Bresser M, Raber F, Klimkait T, Battegay M, Glass TR, Labhardt ND. Offering ART refill through community health workers versus clinic-based follow-up after home-based same-day ART initiation in rural Lesotho: The VIBRA cluster-randomized clinical trial. PLoS Med. 2021 Oct 21;18(10):e1003839. doi: 10.1371/journal.pmed.1003839. eCollection 2021 Oct. PMID 34673765
- [Derived] Amstutz A, Lejone TI, Khesa L, Muhairwe J, Nsakala BL, Tlali K, Bresser M, Tediosi F, Kopo M, Kao M, Klimkait T, Battegay M, Glass TR, Labhardt ND. VIBRA trial - Effect of village-based refill of ART following home-based same-day ART initiation vs clinic-based ART refill on viral suppression among individuals living with HIV: protocol of a cluster-randomized clinical trial in rural Lesotho. Trials. 2019 Aug 22;20(1):522. doi: 10.1186/s13063-019-3510-5. PMID 31439004
- See also: Official Project Website — https://getonproject.wordpress.com

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol V6 approved by Ethics Board on May 30, 2018 (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03630549/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Amended Protocol V7 approved by Ethics Board on Oct 9, 2018 (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03630549/Prot_SAP_003.pdf